CLINICAL TRIAL: NCT01445145
Title: An Exploratory Study of the Use of Five Wishes as a Tool for Advanced Care Planning in Young Adults With Metastatic, Recurrent, or Progressive Cancer or HIV Infection
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070085; 07-C-0085; NCT00445640 (obsolete NCT alias)
Record Dates: First submitted 2011-09-30; First posted 2011-10-03 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2014-09-25

CONDITIONS: Neoplasms
Keywords: End-of-Life; Advance Directive; Pediatric Cancer; Adolescents; Young Adults
MeSH Terms: conditions — Neoplasms; Death

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Few resources exist for helping adolescents and young adults with cancer or HIV disease understand their changing physical, emotional and social needs when treatment is no longer effective.
* An advance directive document called Five Wishes has had particular success with the adult population because of the consideration of personal, emotional and spiritual needs in addition to medical and legal concerns.

Objectives:

-To learn which questions in Five Wishes are useful for adolescents and young adults and to then create a new document that reflects the issues they feel are most appropriate for people with cancer or HIV disease.

Eligibility:

-Adolescents and young adults 16 to 30 years of age with advanced cancer or HIV disease acquired perinatally or early in life and enrolled in an active NIH treatment protocol.

Design:

* Stage 1: Participants go through each question in Five Wishes and respond to whether they feel the questions are useful.
* Stage 2: Participants are asked to compare each question from Five Wishes to a newly developed document based on the feedback received during first stage of the study.
* Participants are enrolled for either Stage 1 or Stage 2 depending on the date they enter the study.

DETAILED DESCRIPTION:
Background:

* Discussing end of life (EoL) care with adolescents and young adults can be one of the most difficult aspects of living with a life threatening disease.
* Few established resources exist to aid this population in accepting and understanding their changing physical, emotional and social needs when treatment is no longer effective. Standards in palliative care suggest that discussion of end of life issues be routine and commence soon after diagnosis.
* While many helpful documents exist to facilitate such conversations with adults, few address the particular concerns and needs of adolescents and young adults.
* One advance directive (AD) document, Five Wishes, has had particular success with the adult population because of the consideration of 'personal, emotional and spiritual needs' in addition to medical and legal concerns.

Objective:

* To determine if adolescents and young adults living with advanced cancer or HIV disease feel that an AD document, such as Five Wishes, is useful in addressing end of life issues.
* To develop and perform a pilot evaluation of a modified age-appropriate advance care planning tool for young adults and adolescents based on Five Wishes that reflects the participants opinions on which questions they feel are most useful and additional items that might be helpful.

Eligibility:

* Age: 16 to 30 years
* Known metastatic, progressive or recurrent cancer or HIV disease acquired perinatally or early in life and enrolled in an active NIH treatment protocol.

Design:

-A descriptive study of attitudes of young adults (16-30 years) with cancer or HIV disease concerning the questions contained in the AD document Five Wishes as well as a comparison between Five Wishes and a modified version of that document.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age: 16 to 30 years
* Patients at NIH or participating site must have 1) a diagnosis of metastatic, recurrent, or progressive cancer with a mean survival rate of 2 years or less or 2) a diagnosis of perinatal or early life transfusion associated HIV infection. The treatment protocol PI or attending physician must consent to have a patient entered into this protocol. Newly diagnosed patients must have completed at least three cycles of chemotherapy.
* For patients less than 18 years of age, a legal guardian must provide informed consent and the patients must sign an assent document.
* Patients greater than 18 years of age must give informed consent.
* Patients less than 18 years of age must have a score of 40 or higher on Lanksy/Karnofsky, as determined by the medical team at the time of enrollment.
* Patients greater than 18 years of age must have a score of 3 or less on the Eastern Cooperative Oncology Group Performance Status Scale (ECOG PS) at the time of enrollment.
* Patients must be English or Spanish speaking.

EXCLUSION CRITERIA:

* Presence of psychotic symptoms or severe psychological distress, which in the judgment of the Principal or Associate Investigator, or consulting psychiatrist would compromise the patient s ability to engage in the intervention or is likely to interfere with the study procedures or results.
* Previously identified cognitive impairment which in the judgment of the Principal or Associate Investigator would compromise the patient s ability to understand the Five Wishes material or is likely to interfere with the study procedures or results.
* Clinically significant, systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction) which in the judgment of the research team would compromise the patient s ability to tolerate this study

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2007-01-26; Study Completion 2014-09-25

CONTACTS AND LOCATIONS:
Overall Officials: Lori Wiener, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Georgetown University, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Wolfe J, Grier HE, Klar N, Levin SB, Ellenbogen JM, Salem-Schatz S, Emanuel EJ, Weeks JC. Symptoms and suffering at the end of life in children with cancer. N Engl J Med. 2000 Feb 3;342(5):326-33. doi: 10.1056/NEJM200002033420506. PMID 10655532
- [Background] Mack JW, Wolfe J. Early integration of pediatric palliative care: for some children, palliative care starts at diagnosis. Curr Opin Pediatr. 2006 Feb;18(1):10-4. doi: 10.1097/01.mop.0000193266.86129.47. PMID 16470155
- [Background] Hammes BJ, Klevan J, Kempf M, Williams MS. Pediatric advance care planning. J Palliat Med. 2005 Aug;8(4):766-73. doi: 10.1089/jpm.2005.8.766. PMID 16128650